CLINICAL TRIAL: NCT01199068
Title: Phase 1b Study of CS-7017 in Combination With Erlotinib in Subjects With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer (NSCLC) Who Failed First-line Therapy
Brief Title: CS-7017 in Combination With Erlotinib in Subjects With Stage IIIb/IV Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS7017-A-A110
Record Dates: First submitted 2010-08-30; First posted 2010-09-10 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: PPAR gamma agonist; Tumor; Cancer; Antineoplastic Agent; Respiratory Tract Neoplasms; Erlotinib; Protein Kinase Inhibitors; Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Respiratory Tract Neoplasms | interventions — efatutazone; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS-7017+Erlotinib (Experimental): Drug: CS-7017 from 0.25 mg to 0.50 mg twice a daily Drug: Erlotinib 150 mg once daily
  Interventions: Drug: CS-7017; Drug: Erlotinib

INTERVENTIONS:
Drug: CS-7017 — CS-7017 from 0.25 mg to 0.50 mg twice daily
  Other Names: CS7017
Drug: Erlotinib — Erlotinib 150 mg once daily
  Other Names: Tarceva

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of CS-7017 administered orally twice a day in combination with erlotinib, and to assess the pharmacokinetics of CS-7017 in combination with erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable locally advanced or metastatic (stage IIIb or IV) Non-small Cell Lung Cancer (NSCLC)
* Recurrent disease (either no response to treatment or subsequent relapse after an objective response) that has progressed after first-line platinum based therapy
* Male or female ≥ 18 years of age
* Anticipation of more than 3 months survival
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 1
* Adequate organ and bone marrow function

Exclusion Criteria:

* Prior Tyrosine Kinase Inhibitor (TKI) therapy
* Anticipation of need for a major surgical procedure or radiation therapy during the study
* Remaining influence of previous therapies such as radiotherapy, surgery, immunotherapy within 4 weeks prior to start of study treatment
* Treatment with anticancer medication within 4 weeks before study treatment, currently enrolled in another investigational drug study, or enrolled in another investigational drug study within 4 weeks of start of treatment
* History of any of the following events within 6 months prior to start of study treatment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class ≥I Congestive Heart Failure (CHF), cerebrovascular accident or cerebral infarction, pulmonary embolism, deep vein thrombosis, or other clinically significant thromboembolic event; clinically significant pulmonary disease (eg, severe Chronic-Obstructive Pulmonary Disease (COPD) or asthma)
* Severe edema, ascites fluid, pericardial or pleural effusion or pericardial involvement with the tumor within 6 months prior to start of study treatment, or which require steroid therapy/ diuretic therapy
* Subjects with brain metastasis (defined as untreated, symptomatic or requiring steroids or anticonvulsant medications to control associated symptoms)
* Subjects with clinically significant active infection which requires antibiotic therapy, or who are hepatitis B surface antigen (HBsAg)-, hepatitis C virus (HCV)- or human immunodeficiency virus (HIV)-positive or receiving antiretroviral therapy
* Subjects with malabsorption syndrome, chronic diarrhea (lasting over 4 weeks), inflammatory bowel disease, or partial bowel obstruction
* Diabetes mellitus requiring insulin, or a history of poor serum glucose control with the use of non-insulin diabetes medications
* Treatment with Thiazolidinedione(TZDs) within 4 weeks prior to start of study treatment
* History of a second malignancy, with the exception of in situ cervical cancer or adequately treated basal cell or squamous cell carcinoma of the skin
* Poorly-controlled blood pressure as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Asan Medical Center, Seoul, Songpa-Gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 participants who met all inclusion and no exclusion criteria were enrolled in the study. Fourteen participants received treatment.
Pre-assignment Details: This study consisted of 2 parts: initial portion and additional portion. In the initial portion, participants received CS-7017 (starting dose 0.25 mg BID ascending to 0.50 mg BID) in combination with erlotinib. In the additional portion, participants received CS-7017 0.50 mg BID in combination with erlotinib.
Groups:
- CS-7017 0.25 mg BID; Initial Portion: Participants who received oral CS-7017 0.25 mg twice daily (BID) in combination with erlotinib 150 mg administered once daily.
- CS-7017 0.50 mg BID; Initial Portion; CS-7017 0.50 mg BID; Additional Portion: Participants who received oral CS-7017 0.50 mg twice daily (BID) in combination with erlotinib 150 mg administered once daily.
Period: Overall Study
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion
Started | 3 | 3 | 9
Received Treatment | 3 | 3 | 8
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 9
Not completed — Unacceptable toxicity | 0 | 0 | 2
Not completed — Progressive disease | 3 | 3 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for participants in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion | Total
Number analyzed (Participants) | 3 | 3 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 7 | 13
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (8.39) | 53.3 (4.04) | 60.0 (9.89) | 57.4 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 4
  Male | 3 | 2 | 5 | 10
Region of Enrollment [Number; unit: participants]
  South Korea | 3 | 3 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: CS-7017-Related Treatment-Emergent Adverse Events Occurring During the Study of Administration of CS-7017 Combined With Erlotinib in Participants With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer Who Failed First-line Therapy
Description: A treatment-emergent adverse event (TEAE) is defined as any event not present prior to the initiation of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment. A CS-7017-related TEAE is an TEAE that is related to CS7017 in the relationship.
Time Frame: From post first dose to 30 days after last dose, up to approximately 1.5 years
Population: CS-7017-related TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- CS-7017 0.50 mg BID; Initial + Additional Portions: Participants who received oral CS-7017 0.50 mg twice daily (BID) in combination with erlotinib 150 mg administered once daily (combined initial and additional portions).
- Overall: All participants who received CS-71017 in combination with erlotinib.
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion | CS-7017 0.50 mg BID; Initial + Additional Portions | Overall
Number analyzed (Participants) | 3 | 3 | 8 | 11 | 14
Participants
  At least one CS-7017-Relaed TEAE | 2 | 2 | 8 | 10 | 12
  Blood and Lymphatic System Disorders | 1 | 1 | 4 | 5 | 6
  Anaemia | 0 | 1 | 4 | 5 | 5
  Thrombocytopenia | 1 | 0 | 1 | 1 | 2
  Neutropenia | 1 | 0 | 0 | 0 | 1
  Metabolism and Nutrition Disorders | 0 | 0 | 5 | 5 | 5
  Decreased appetite | 0 | 0 | 4 | 4 | 4
  Hypokalaemia | 0 | 0 | 1 | 1 | 1
  Hyponatraemia | 0 | 0 | 1 | 1 | 1
  Eye Disorders | 0 | 0 | 1 | 1 | 1
  Conjunctival hyperaemia | 0 | 0 | 1 | 1 | 1
  Cardiac Disorders | 0 | 0 | 3 | 3 | 3
  Pericardial effusion | 0 | 0 | 3 | 3 | 3
  Sinus arrhythmia | 0 | 0 | 1 | 1 | 1
  Respiratory, Thoracic, and Mediastinal Disorders | 0 | 0 | 3 | 3 | 3
  Pleural effusion | 0 | 0 | 3 | 3 | 3
  Gastrointestinal Disorders | 0 | 0 | 2 | 2 | 2
  Nausea | 0 | 0 | 2 | 2 | 2
  Renal and Urinary Disorders | 0 | 0 | 1 | 1 | 1
  Azotaemia | 0 | 0 | 1 | 1 | 1
  Congenital, Familial, and Genetic Disorders | 0 | 1 | 0 | 1 | 1
  Hydrocele | 0 | 1 | 0 | 1 | 1
  General Disorders & Administration Site Conditions | 2 | 1 | 8 | 9 | 11
  Face oedema | 2 | 1 | 8 | 9 | 11
  Oedema peripheral | 1 | 1 | 5 | 6 | 7
  Fatigue | 0 | 0 | 2 | 2 | 2
  Generalised oedema | 0 | 0 | 2 | 2 | 2
  Malaise | 0 | 0 | 1 | 1 | 1
  Investigations | 1 | 1 | 7 | 8 | 9
  Weight increased | 1 | 1 | 7 | 8 | 9
  Blood creatinine increased | 0 | 0 | 2 | 2 | 2
  Blood creatinine phosphokinase increased | 0 | 0 | 1 | 1 | 1
  Brain natriuretic peptide increased | 0 | 0 | 1 | 1 | 1
  Electrocardiogram QT prolonged | 0 | 0 | 1 | 1 | 1

2. Primary Outcome: Pharmacokinetic Parameter Area Under the Concentration Versus Time Curve of Serum Free Form of CS-7017 (R-150033) After CS-7017 and Erlotinib in Participants With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer
Description: After the first CS-7017 administration, area under the concentration-time curve from zero to the last quantifiable concentration (AUClast) and area under the concentration-time curve during dosing interval (AUCtau) were assessed.
Time Frame: Cycle 1, Week 1 and Cycle 2, Week 4
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial + Additional Portions
Number analyzed (Participants) | 3 | 11
ng*h/mL
  Cycle 1, Week 1: AUClast | 50.8 (38.6) | 148 (84.3)
  Cycle 1, Week 1: AUCtau: number analyzed (Participants) | 2 | 11
  Cycle 1, Week 1: AUCtau | 97.2 (45.8) | 205 (115)
  Cycle 2, Week 4: AUClast: number analyzed (Participants) | 2 | 7
  Cycle 2, Week 4: AUClast | 124 (22.8) | 212 (104)
  Cycle 2, Week 4: AUCtau: number analyzed (Participants) | 2 | 7
  Cycle 2, Week 4: AUCtau | 174 (27.0) | 307 (156)

3. Primary Outcome: Pharmacokinetic Parameter Observed Serum Concentration (Cmax) of Serum Free Form of CS-7017 (R-150033) After CS-7017 and Erlotinib in Participants With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer
Description: After the first CS-7017 administration, observed serum concentration (Cmax) and observed serum concentration at steady state (Cmax,ss) were assessed.
Time Frame: Cycle 1, Week 1 and Cycle 2, Week 4
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial + Additional Portions
Number analyzed (Participants) | 3 | 11
ng/mL
  Cycle 1, Week 1: Cmax | 9.98 (6.20) | 25.1 (14.0)
  Cycle 2, Week 4: Cmax,ss: number analyzed (Participants) | 2 | 7
  Cycle 2, Week 4: Cmax,ss | 18.9 (3.75) | 32.4 (16.0)

4. Primary Outcome: Pharmacokinetic Parameter Time of Maximum Plasma Concentration (Tmax) of Serum Free Form of CS-7017 (R-150033) After CS-7017 and Erlotinib in Participants With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer
Description: After the first CS-7017 administration, time of maximum plasma concentration (Tmax) and time of maximum plasma concentration at steady state (Tmax,ss) were assessed.
Time Frame: Cycle 1, Week 1 and Cycle 2, Week 4
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: h
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial + Additional Portions
Number analyzed (Participants) | 3 | 11
h
  Cycle 1, Week 1: Tmax | 3.00 [2.00 to 8.00] | 3.00 [1.95 to 4.00]
  Cycle 2, Week 4: Tmax,ss: number analyzed (Participants) | 2 | 7
  Cycle 2, Week 4: Tmax,ss | 3.50 [3.00 to 4.00] | 3.00 [0.50 to 4.02]

5. Secondary Outcome: Best Overall Response and Response Rate Following Administration of CS-7017 in Combination With Erlotinib in Participants With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer (NSCLC) Who Failed First-line Therapy
Description: As per Response Evaluation Criteria for Solid Tumors v1.1, best overall response was characterized as complete response (CR) defined as disappearance of all target lesions, partial response (PR) defined as
  ≥30% decrease in the sum of diameters of target lesions, progressive disease (PD) defined as ≥20% increase in the sum of diameters of target lesions, and stable disease (SD) defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Response rate was defined as CR + PR.
Time Frame: From screening and after completion of every 2 cycles (6 weeks) until disease progression, withdrawal of consent, death, or loss to follow-up, up to approximately 1.5 years
Population: Best overall response and response rate were assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion | CS-7017 0.50 mg BID; Initial + Additional Portions | Overall
Number analyzed (Participants) | 2 | 3 | 7 | 10 | 12
Participants
  Partial response (PR) | 0 | 0 | 5 | 5 | 5
  Stable disease (SD) | 2 | 1 | 1 | 2 | 4
  Progressive disesae (PD) | 0 | 2 | 1 | 3 | 3
  Response rate (CR+PR) | 0 | 0 | 5 | 5 | 5

6. Secondary Outcome: Progression-free Survival Time Following Administration of CS-7017 in Combination With Erlotinib in Participants With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer (NSCLC) Who Failed First-line Therapy
Description: Progression-free survival (PFS) was defined as the time from randomization to the date of the first objective documentation of progressive disease (PD) or death resulting from any cause, whichever came first.
Time Frame: From randomization to PD or death, up to approximately 1.5 years
Population: Per-protocol Progression-free Survival Time data was only assessed in the 0.50 mg BID (additional portion) and the 0.5 mg BID (initial and additional portions) Groups.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CS-7017 0.50 mg BID; Additional Portion | CS-7017 0.50 mg BID; Initial + Additional Portions | Overall
Number analyzed (Participants) | 7 | 10 | 12
days | 125 [82 to 176] | 82 [41 to 176] | 84 [64 to 127]

7. Secondary Outcome: Erlotinib-Related Treatment-Emergent Adverse Events Occurring During the Study of Administration of CS-7017 Combined With Erlotinib in Participants With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer Who Failed First-line Therapy
Description: A treatment-emergent adverse event (TEAE) is defined as any event not present prior to the initiation of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment. An erlotinib-related TEAE is an TEAE that is related to erlotinib in the relationship
Time Frame: From post first dose to 30 days after last dose, up to approximately 1.5 years
Population: Erlotinib-related TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion | CS-7017 0.50 mg BID; Initial + Additional Portions | Overall
Number analyzed (Participants) | 3 | 3 | 8 | 11 | 14
Participants
  At least one erolitinib-related TEAE | 3 | 3 | 8 | 11 | 14
  Infections and Infestations | 1 | 0 | 1 | 1 | 2
  Paronychia | 1 | 0 | 1 | 1 | 2
  Blood and Lymphatic System Disorders | 0 | 0 | 1 | 1 | 1
  Anaemia | 0 | 0 | 1 | 1 | 1
  Metabolism and Nutrition Disorders | 0 | 0 | 4 | 4 | 4
  Decreased appetite | 0 | 0 | 4 | 4 | 4
  Eye Disorders | 0 | 0 | 3 | 3 | 3
  Blepharitis | 0 | 0 | 1 | 1 | 1
  Conjunctival hyperaemia | 0 | 0 | 1 | 1 | 1
  Dry eye | 0 | 0 | 1 | 1 | 1
  Respiratory, Thoracic, and Mediastinal Disorders | 0 | 1 | 2 | 3 | 3
  Nasal dryness | 0 | 0 | 1 | 1 | 1
  Nasal inflammation | 0 | 1 | 0 | 1 | 1
  Oropharyngeal pain | 0 | 0 | 1 | 1 | 1
  Gastrointestinal Disorders | 1 | 2 | 8 | 10 | 11
  Diarrhoea | 1 | 2 | 6 | 8 | 9
  Nausea | 0 | 0 | 2 | 2 | 2
  Anorectal discomfort | 0 | 1 | 0 | 1 | 1
  Flatulence | 0 | 0 | 1 | 1 | 1
  Stomatitis | 0 | 0 | 1 | 1 | 1
  Skin and Subcutaneous Tissue Disorders | 3 | 2 | 8 | 10 | 13
  Skin exfoliation | 2 | 1 | 6 | 7 | 9
  Dry skin | 2 | 1 | 5 | 6 | 8
  Rash | 0 | 0 | 7 | 7 | 7
  Dermatitis acneiform | 3 | 2 | 1 | 3 | 6
  Pruritus | 2 | 1 | 3 | 4 | 6
  Alopecia | 0 | 0 | 1 | 1 | 1
  Renal and Urinary Disorders | 0 | 0 | 1 | 1 | 1
  Azotaemia | 0 | 0 | 1 | 1 | 1
  General Disorders & Administration Site Conditions | 0 | 0 | 2 | 2 | 2
  Fatigue | 0 | 0 | 2 | 2 | 2
  Investigations | 0 | 0 | 2 | 2 | 2
  Blood creatinine increased | 0 | 0 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event data were collected from after the first dose up to 30 days after the last dose, up to approximately 1.5 years in the Safety Analysis Set.
Description: Adverse events (AEs) were defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All-cause mortality includes all deaths that occurred during the study and within 30 days after the last dose of study drug.
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion | CS-7017 0.50 mg BID; Initial + Additional Portions | Overall
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 0/8 | 1/11 | 2/14
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 4/8 | 7/11 | 8/14
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 8/8 | 11/11 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 0.25 mg BID; Initial Portion (N=3) | CS-7017 0.50 mg BID; Initial Portion (N=3) | CS-7017 0.50 mg BID; Additional Portion (N=8) | CS-7017 0.50 mg BID; Initial + Additional Portions (N=11) | Overall (N=14)
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 2 | 2
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 0.25 mg BID; Initial Portion (N=3) | CS-7017 0.50 mg BID; Initial Portion (N=3) | CS-7017 0.50 mg BID; Additional Portion (N=8) | CS-7017 0.50 mg BID; Initial + Additional Portions (N=11) | Overall (N=14)
Paronychia (Infections and infestations) | 1 | 0 | 1 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 2 | 2
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 5 | 7 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 6 | 8 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 4 | 5 | 5
Headache (Nervous system disorders) | 0 | 1 | 1 | 2 | 2
Depressed level of consciousness (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1 | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 1 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 3 | 3 | 3
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2 | 2 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 7 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4 | 7 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 2
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 6 | 8 | 9
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 3 | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2 | 4 | 4
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 4 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 3
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastritis atropic (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 1 | 6 | 7 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 5 | 6 | 8
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 7 | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 3 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 4 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 4 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1 | 1
Face oedema (General disorders) | 2 | 1 | 8 | 9 | 11
Oedema peripheral (General disorders) | 1 | 2 | 5 | 7 | 8
Fatigue (General disorders) | 1 | 1 | 3 | 4 | 5
Asthenia (General disorders) | 1 | 1 | 2 | 3 | 4
Generalised oedema (General disorders) | 0 | 0 | 2 | 2 | 2
Chest discomfort (General disorders) | 0 | 0 | 1 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 1 | 1 | 1
Puncture site pain (General disorders) | 0 | 0 | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 1
Weight increased (Investigations) | 2 | 1 | 7 | 8 | 10
Blood creatinine phosphokinase increased (Investigations) | 2 | 0 | 1 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 2 | 2
Weight decreased (Investigations) | 0 | 0 | 2 | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 1 | 1
Electrocardiogram QC prolonged (Investigations) | 0 | 0 | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No